CLINICAL TRIAL: NCT01150448
Title: An Open-Label, Long-Term, Multiple-Dose, Safety and Tolerability, Pharmacokinetic Study of 150 mg eq. Paliperidone Palmitate in the Treatment of Subjects With Schizophrenia
Brief Title: A Safety and Pharmacokinetic Study of Paliperidone Palmitate in Patients With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CR013300; R092670PSY1008
Record Dates: First submitted 2010-06-17; First posted 2010-06-25 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Schizophrenia
Keywords: Paliperidone palmitate; paliperidone ER (INVEGA); R092670PSY1008; Risperidone; Risperdal (RISPERDAL CONSTA); Pharmacokinetics
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 001 (Experimental): Paliperidone palmitate Treatment A All patients will receive a single IM injection of 150mg eq of study drug on Day 1. Patients who tolerate 150mg eq will receive a 2nd IM injection of 150mg eq on Day 8 followed by 12 IM injections (1 every 4 weeks) of 150mg eq. All other patients will be assigned to Treatment B.
  Interventions: Drug: Paliperidone palmitate Treatment A
- 002 (Experimental): Paliperidone palmitate Treatment B Patients not tolerating Treatment A will receive a single IM injection of study drug 100mg eq at their next scheduled visit followed by injections (1 every 4 weeks) ranging from 50 to 150mg eq patients who do not wish to have multiple blood samples collected will also be assigned to Treatment B
  Interventions: Drug: Paliperidone palmitate Treatment B

INTERVENTIONS:
Drug: Paliperidone palmitate Treatment A — All patients will receive a single IM injection of 150mg eq of study drug on Day 1. Patients who tolerate 150mg eq will receive a 2nd IM injection of 150mg eq on Day 8 followed by 12 IM injections (1 every 4 weeks) of 150mg eq. All other patients will be assigned to Treatment B.
  Arms: 001
Drug: Paliperidone palmitate Treatment B — Patients not tolerating Treatment A will receive a single IM injection of study drug 100mg eq at their next scheduled visit followed by injections (1 every 4 weeks) ranging from 50 to 150mg eq
  Arms: 002

SUMMARY:
The purpose of this study is to evaluate the long term safety of flexible doses (50 to 150 mg equivalent) of paliperidone palmitate in the treatment of patients with schizophrenia and to document the pharmacokinetics of paliperidone following fixed multiple intramuscular injections of paliperidone palmitate 150 mg eq.

DETAILED DESCRIPTION:
This is an open-label (identity and dose of study drug will be known to patients), safety and pharmacokinetic study of the highest dose (150 mg equivalent) of paliperidone palmitate (referred to as study drug) administered by intramuscular (IM) injection (injection into the muscle) in patients with schizophrenia. A total of at least 200 adult patients with schizophrenia will participate in the study. The study will consist of 2 phases: an up-to-21-day screening period and a 53-week open-label treatment period including an end of study/withdrawal visit. The total duration of the study will be approximately 56 weeks. At the screening visit, if a patient has been treated with an antipsychotic medication before study entry, the medication may be continued during the study except for protocol-specified medications that are not permitted. If patients have not received previous treatment with at least 2 oral (by mouth) doses of the antipsychotic agents risperidone or paliperidone or 1 dose of injectable RISPERDAL CONSTA or paliperidone palmitate, they will undergo a 4-day evaluation period and receive a 6 mg/day oral dose of an extended-release (ER) formulation of paliperidone to evaluate their ability to tolerate study drug. Patients who are able to tolerate study drug and meet all other entry criteria for the study will then be administered a single IM injection into the deltoid muscle (upper arm) of paliperidone palmitate 150 mg equivalent (eq) on Day 1 (Treatment A). Patients who tolerate Treatment A will receive a 2nd IM injection in the deltoid muscle of 150 mg eq on Day 8 followed by 150 mg eq administered by IM injection in the deltoid or gluteal (buttocks) muscle once every 4 weeks for the remainder of the 53-week treatment period. Patients who do not tolerate Treatment A or who do not wish to have multiple blood samples collected for pharmacokinetic testing will be assigned to Treatment B. Patients who do not tolerate Treatment A will receive a single IM injection of study drug 100 mg eq at their next scheduled visit followed by a flexible dose schedule of study drug ranging from 50 to 150 mg eq administered by IM injection in the deltoid or gluteal muscle every 4 weeks for the remainder of the 53-week treatment period. Blood samples for pharmacokinetics (ie, to test the concentration of study drug in the blood) will be collected at specified times before and after each dose of study drug from all patients; additional blood samples for pharmacokinetic testing will be collected from patients receiving Treatment A. An additional blood sample may also be collected at any time during screening or before the first day of IM administration of study drug for patients who agree to participate in an optional part of the study called a pharmacogenomic evaluation (genetic testing) for possible use in characterizing the safety and/or efficacy of study drug in relation to the pharmacogenic (genetic) profile of the patient. Periodically during the study, patients will be assessed for the presence of psychiatric symptoms and severity of symptoms. The safety and tolerability of paliperidone will be evaluated by monitoring adverse events (side effects) and relevant changes in laboratory values, electrocardiogram (ECG), vital signs measurements, physical examinations, and extrapyramidal symptoms (ie, symptoms that can be associated with taking antipsychotic drugs) scores reported from the time of screening to the end of the study (Day 372 or at the time of the patient's early termination from the study). The concentration of paliperidone in plasma (colorless portion of blood) from blood samples collected from Day 1 through to the end of the study will also be determined. Since only limited information exists regarding the repeated administration of doses of paliperidone palmitate, an internal review board will meet 2 times during the study to review safety data collected. The first review of safety data will be performed after approximately 30 patients complete 99 days of treatment and the second review of safety data will be made after approximately 75 patients complete 176 days of treatment. After each review of safety data, the safety review board will make a recommendation to continue the study, modify the protocol, or to terminate the study. Patients will receive 1 injection in the deltoid muscle of Treatment (Tx) A (study drug 150mg eq) on Day 1. Patients will then receive 1 injection in the deltoid muscle of Tx A on Day 8 followed by 1 injection every 4 weeks in the deltoid or gluteal muscle OR patients will be assigned to Txt B and receive 1 injection in the deltoid or gluteal muscle of study drug 100mg eq at next visit followed by 1 injection every 4 weeks of study drug 50 to 150mg eq in the deltoid or gluteal muscle.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) for at least 1 year before screening
* Have a body mass index (BMI) of >=17.0 kg/m2 at screening
* Have a Positive and Negative Syndrome Scale (PANSS) total score of <=70

Exclusion Criteria:

* Have a primary active DSM-IV Axis I diagnosis other than schizophrenia
* Have a PANSS total score of >70 at screening
* Have a PANSS score of >16 points on the sum of the following 4 items at screening and baseline: conceptual disorganization, suspiciousness/persecution, hallucinatory behavior, and unusual thought content
* Have scores greater than 5 on any of the individual items of the PANSS at screening or baseline
* Have attempted suicide within 12 months before screening or are at imminent risk of suicide or violent behavior as clinically assessed by the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2007-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The number of patients experiencing treatment emergent adverse events | Screening (Day -21 to -1) to Day 372 (or at the time of early termination from the study)
Concentration of paliperidone in plasma from blood samples obtained from patients | Day 1 to Day 372

SECONDARY OUTCOMES:
Changes in Sleep Visual Analog Scale (Sleep VAS) scores as an indicator of quality of sleep and daytime drowsiness | Day 1 to Day 372.
Changes in Positive and Negative Syndrome Scale (PANSS) scores | Day 1 to Day 372.
Change in Clinical Global Impression Severity of Illness (CGI-S) Scores as an indicator of overall clinical condition | Day 1 to Day 372.
Changes in Personal and Social Performance Scale (PSP) Scores (measures personal and social performance in patients with acute symptoms of schizophrenia. Higher PSP scores indicate better personal and social functioning) | Day 1 to Day 372.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (28):
- United States (5):
  - Cerritos, California
  - National City, California
  - San Diego, California
  - Atlanta, Georgia
  - Philadelphia, Pennsylvania
- Aalst, Belgium
- Zagreb, Croatia
- Kuala Lumpur, Malaysia
- Poland (4):
  - Leszno
  - Lubliniec
  - Poznan
  - Torun
- Slovakia (3):
  - Bratislava
  - Michalovce
  - Rimavská Sobota
- South Korea (3):
  - Gwangju
  - Incheon
  - Seoul
- Spain (3):
  - Badalona
  - Barcelona
  - Madrid
- Taiwan (5):
  - Hualien City
  - Kaohsiung City
  - Tainan
  - Taipei
  - Taoyuan District
- Thailand (2):
  - Bangkok
  - Chiang Mai

REFERENCES:
- [Derived] Coppola D, Liu Y, Gopal S, Remmerie B, Samtani MN, Hough DW, Nuamah I, Sulaiman A, Pandina G. A one-year prospective study of the safety, tolerability and pharmacokinetics of the highest available dose of paliperidone palmitate in patients with schizophrenia. BMC Psychiatry. 2012 Mar 28;12:26. doi: 10.1186/1471-244X-12-26. PMID 22455454
- See also: A Safety and Pharmacokinetic Study of Paliperidone Palmitate in Patients with Schizophrenia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=759&filename=CR013300_CSR.pdf
- See also: A Safety and Pharmacokinetic Study of Paliperidone Palmitate in Patients with Schizophrenia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=759&filename=CR013300_JNL1.pdf